CLINICAL TRIAL: NCT05945420
Title: Outcome of Adding Desmopressin to Tamsulosin for Treatment of Nocturnal Polyurea in Patients With Benign Prostatic Obstruction
Brief Title: Adding Desmopressin to Tamsulosin for Treatment of BPH
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MS.22.12.2245
Record Dates: First submitted 2023-05-31; First posted 2023-07-14 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Nocturnal Polyurea in Patients With BPH
MeSH Terms: interventions — Deamino Arginine Vasopressin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Desmopressin arm (Active Comparator): This arm will receive tamsulosin and desmopressin
  Interventions: Drug: Desmopressin Acetate
- Placebo arm (Placebo Comparator): This arm will receive tamsulosin and placepo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Desmopressin Acetate — This arm will receive tamsulosin and desmopressin acetate daily a
  Arms: Desmopressin arm
Drug: Placebo — This arm will receive tamsulosin and placebo
  Arms: Placebo arm

SUMMARY:
In this study investigators will add desmopressin for treatment of patients with benign prostatic hyperplasia and nocturnal polyurea

DETAILED DESCRIPTION:
Investigators will give a group of patients tamsulosin and desmopressin and the other group will take tamsulosin and placepo and compare the outcome regarding symptoms of being prostatic hyperplasia especially nocturia and the effect on nocturnal polyurea in patients

ELIGIBILITY:
Inclusion Criteria:

Men with BPH Age more than 50years Patients with nocturia (2voids per night or More) Patients with nocturnal polyurea (urine volume More than 33%of urine allover the day) IPSS more than 12 Obstructed flow curve Post voiding residual less than 150

Exclusion Criteria:

* men with BPH with : Acute urine retention Neurogenic bladder dysfunction Cardiovascular disease Hyponatremia Urethral stricture Bladder calculi Prostate cancer

Ages: 50 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2023-07-20 (Estimated); Primary Completion 2024-01-10 (Estimated); Study Completion 2024-02-10 (Estimated)

PRIMARY OUTCOMES:
Change of symptoms and nocturia disappears or improve | Follow up for 6 months
  Investigators will compare symptoms in the pretreatment period and follow up symptoms following treatment and record the outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Urology and nephrology center, Al Mansurah, Outside U.S./Canada, Egypt